CLINICAL TRIAL: NCT06730139
Title: Oral Health Related Quality of Life in Head and Neck Cancer Survivors Within the First Year Following Treatment: a Cross Sectional Study in Egypt
Brief Title: Oral Health Related Quality of Life in Head and Neck Cancer Survivors Within the First Year Following Treatment
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma ElSayed, assistant professor of Oral Medicine, Periodontology, and Oral Diagnosis, Faculty of Dentistry, King Salman International University, El-tor, Egypt., Ain Shams University
Other Study IDs: MAM00213
Record Dates: First submitted 2024-12-06; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer (HNC); Oral Health-Related Quality of Life (OHRQoL); Radiation Therapy (RT); Oral Complications; Quality of Life
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Head and Neck Cancer (HNC) Survivors: Target Population:
  Age: 18 years and older Diagnosis: Head and Neck Cancer (HNC) Treatment Status: Within the first year post-treatment completion

SUMMARY:
Oral Health-Related Quality of Life in Head and Neck Cancer Patients

Problem Statement:

Head and Neck Cancer (HNC) is a significant global health issue, and its incidence is rising. While treatment options have improved, they often lead to severe oral complications, impacting patients' quality of life.

Research Gap:

Limited research exists on oral health-related quality of life (OHRQoL) among HNC patients in Egypt, particularly focusing on the impact of oral clinical parameters and treatment-related factors.

Research Objective:

To assess the OHRQoL of HNC patients who have completed treatment within the past 12 months and to identify factors associated with impaired OHRQoL.

Methodology:

This study will employ a comprehensive approach to evaluate OHRQoL, considering:

Oral Clinical Parameters: Oral hygiene status, oral mucositis, and other oral health indicators.

Sociodemographic Factors: Age, gender, education, occupation, and socioeconomic status.

Treatment-Related Variables: Type of treatment (surgery, radiation therapy, chemotherapy), treatment duration, and dose intensity.

Expected Outcomes:

The findings of this study will:

Quantify the impact of HNC treatment on OHRQoL. Identify key factors associated with impaired OHRQoL. Highlight the importance of standardized oral care for HNC patients. Provide evidence-based recommendations for improving oral health support and enhancing the overall quality of life for HNC survivors.

By addressing the oral health needs of HNC patients, this research aims to improve their quality of life and contribute to better long-term outcomes.

DETAILED DESCRIPTION:
Head and neck cancer (HNC) is the seventh most common cancer globally, accounting for more than 660,000 new cases and 325,000 deaths annually. The number of HNC cases is expected to grow by 30% each year until 2030.[1] The rise has been observed in both developed and developing countries.[2] The survival for HNC has improved modestly over the past three decades with the introduction of different and multi-disciplinary treatment modalities.[3] There are several treatment options for HNC, including radiation therapy, surgery, and chemotherapy. These treatments can be used alone or in combination. Radiation therapy (RT) involves using high-energy beams to destroy cancer cells, while it is an important part of HNC treatment, it can also cause various toxicities, sometimes severe, toxicities.[4].

In most of the cases, head and neck tumors may destroy organs that play an important part in daily activities such as eating and speaking [5]. Additionally, the therapeutic approaches for the treatment of cancer usually result in collateral effects [6]. that impact in the quality of life. The assessment of the quality of life in patients with cancer became a valuable tool to investigate the progression of the disease and the effectiveness of the treatment [7].

The oral condition has an essential role in the individual's systemic health [8]. In specific, the quality of lifer elated to oral health (OHRQoL) may be defined as the lack of negative impact of the oral condition on social, psychological and functional activities [9]. In general, patients with tumors in the oral cavity figure amongst the worst indices for the quality of life when compared to patients with tumors in other regions [10]. Based on the exposed, the present study aimed to measure the impact of OHRQoL of patients with HNC and to evaluate the factors associated.

QoL assessment is an important tool for evaluating not only the impact of disease and its treatment on an individual level but also helpful in developing and revising the rehabilitative ser- vices and patient education material to further improve the clinical outcomes (survival) of patients [11]. Oral health related quality of life (OHRQoL), specifically focuses on self-report aspects pertaining to oral health, capturing the functional, social, and psychological dimensions affected by oral disease [12]. In the case of HNC, disruptions in key oral functions poses a higher risk of adversely affecting both OHRQoL and overall QoL[13].

Not much evidence is found in Egypt related to oral care measures for HNC patients, such as professional care by a dentist and dental hygienist (mechanical or manual removal of mucosal debris, oral hygiene counsel- ling, etc.) at least once a week until the completion of RT [14]. The patients are often unaware of the potential harm from the cancer treatment, only a proportion of HNC patients seek dental consultation for their complications, and most of them suffer greatly even after the completion of treatment due to disturbed oral functions.

To the best of our knowledge, this study represents the first comprehensive assessment of OHRQoL in HNC treated patients who had completed their cancer treatment within the past 12 months. Additionally, it aims to explore the associations between various oral clinical parameters, including oral hygiene status and oral mucositis, and several predictive factors such as sociodemographic characteristics and treatment-related variables in relation to OHRQoL. The findings of this study will highlights the importance of standardizing oral care and improving oral health support for HNC treated patients to reduce the impact of oral problems which can negatively impact their overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Diagnosed with HNC
* Within the first year post-cancer treatment
* Scheduled for a routine follow-up visit at AMTH
* Presence of at least one molar and one central incisor in each jaw
* Able to provide informed consent

Exclusion Criteria:

* Inability to provide informed consent
* Debilitative conditions or cognitive disabilities
* Trismus (mouth opening < 20 mm)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of HNC survivors who meet the following criteria:
  Age: 18 years and older Treatment Completion: Within the past year Dental Status: Presence of at least one molar and one central incisor in the upper and lower jaw Cognitive Function: No cognitive disabilities or debilitating conditions Mouth Opening: Minimum of 20 mm Participants will be recruited from the oncology unit at Ahmed Maher Teaching Hospital (AMTH) during their routine follow-up visits. Eligible patients will be informed about the study and provided with a written informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
European Organization for Treatment of Cancer Quality of Life Questionnaire for Head and Neck Cancer (EORTC QLQ-H&N-35). | Assessed once during the study (day 1 of the study)
  EORTC QLQ-H&N-35 Minimum Score: 0 Maximum Score: 100 Higher Scores: Indicate worse outcomes and more severe symptoms.
  Domains Evaluated:
  Functional Domains:
  Pain and soreness in the mouth and throat
  Swallowing difficulties Taste and smell alterations Social eating and enjoyment of meals Social contact Sexuality
  Symptom Scale:
  Teeth problems Mouth opening difficulties Dry mouth Sticky saliva Coughing Feeling ill Pain killer use
  Nutritional supplement or feeding tube use
  Weight loss
  Weight gain

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Maher teaching hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No